CLINICAL TRIAL: NCT03492463
Title: The Role of Nicotine Dose and Route of Delivery in Affecting Adoption of E-cigarettes and Reducing Exposure to Toxic Combustion Products
Acronym: ENDS-Switch
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00084132; P50DA027840-07 (NIH)
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Nicotine Dependence, Cigarettes
Keywords: Nicotine addiction; Cigarette smoking; Nicotine patches; E-cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Vaping | interventions — Tobacco Use Cessation Devices; Nicotine; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nicotine e-cigs + Nicotine patches (Active Comparator): Participants will receive e-cigarettes containing nicotine and nicotine patches (21mg/24hr) and will be asked to switch from cigarette use to use of the study e-cigarettes for eight weeks.
  Interventions: Drug: Nicotine patch; Other: E-cigarettes
- Non-nicotine e-cigs + Nicotine patches (Active Comparator): Participants will receive e-cigarettes not containing nicotine and nicotine patches (21mg/24hr) and will be asked to switch from cigarette use to use of the study e-cigarettes for eight weeks.
  Interventions: Drug: Nicotine patch; Other: Non-nicotine e-cigarettes
- Nicotine e-cigs + Placebo patches (Active Comparator): Participants will receive e-cigarettes containing nicotine and placebo patches (21mg/24hr) and will be asked to switch from cigarette use to use of the study e-cigarettes for eight weeks.
  Interventions: Other: Placebo patch; Other: E-cigarettes
- Non-nicotine e-cigs + Placebo patches (Placebo Comparator): Participants will receive e-cigarettes not containing nicotine and placebo patches (21mg/24hr) and will be asked to switch from cigarette use to use of the study e-cigarettes for eight weeks.
  Interventions: Other: Placebo patch; Other: Non-nicotine e-cigarettes

INTERVENTIONS:
Drug: Nicotine patch — Participants will wear the nicotine patch daily while switching from cigarette use to use of e-cigarettes for eight weeks.
  Other Names: NicoDerm
  Arms: Nicotine e-cigs + Nicotine patches; Non-nicotine e-cigs + Nicotine patches
Other: Placebo patch — Participants will wear the placebo patch daily while switching from cigarette use to use of e-cigarettes for eight weeks.
  Arms: Nicotine e-cigs + Placebo patches; Non-nicotine e-cigs + Placebo patches
Other: E-cigarettes — Participants will use e-cigarettes containing nicotine while switching from cigarette use to use of e-cigarettes for eight weeks.
  Other Names: Electronic Nicotine Delivery System (ENDS); e-cigs; electronic cigarettes
  Arms: Nicotine e-cigs + Nicotine patches; Nicotine e-cigs + Placebo patches
Other: Non-nicotine e-cigarettes — Participants will use e-cigarettes not containing nicotine while switching from cigarette use to use of e-cigarettes for eight weeks.
  Other Names: Electronic Nicotine Delivery System (ENDS); e-cigs; electronic cigarettes
  Arms: Non-nicotine e-cigs + Nicotine patches; Non-nicotine e-cigs + Placebo patches

SUMMARY:
This study plans to investigate whether using electronic cigarettes (e-cigarettes) or skin patches containing nicotine affects switching from smoking conventional combustible (burning) cigarettes.

DETAILED DESCRIPTION:
This study proposes to assess the relative role of nicotine dose and route of delivery in affecting successful switching from combustible cigarettes to e-cigarettes, as well as concomitant reductions in ad libitum cigarette smoking and exposure to harmful and potentially harmful constituents of combustion. The strategy will be to assess adoption of e-cigarette use and concomitant reduction in ad libitum smoking of subjects' usual brands of cigarettes over an 8-week period, during which they will receive nicotine or non-nicotine e-cigarettes, and nicotine skin patches. The nicotine patches will not be used as a therapeutic treatment in this study, but rather as a way to manipulate the nicotine dose, while varying the rate and route of nicotine delivery. Behavioral or "habit" aspects of e-cigarette use will be controlled for by the groups receiving non-nicotine e-cigarettes. Initially the study design included placebo patch control conditions, but due to limitations in budget and period of support, enrollment in these these arms was discontinued. All participants currently receive active nicotine patches.

ELIGIBILITY:
Inclusion Criteria:

* Smoke an average of at least 10 cigarettes per day;
* Have smoked at least one cumulative year;
* Have an expired air CO reading of at least 10ppm;
* Have a body weight of > 110 lbs. (50 kg) and ≤ 300 lbs. (136 kg);
* Are able to read and understand English;

Potential subjects of child bearing potential must agree to use acceptable contraception during their participation in this study. Potential subjects must agree to avoid the following during their participation in this study:

* Participation in any other nicotine-related modification strategy outside of this protocol;
* Use of tobacco products other than cigarettes, including pipe tobacco, cigars, snuff, and chewing tobacco;
* Use of e-cigarettes other than the ones provided during the study;
* Use of experimental (investigational) drugs or devices;
* Use of illegal drugs;
* Use of exclusionary medications.

Exclusion Criteria:

* Seeking treatment for nicotine dependence.
* Hypertension - systolic BP > 160 mm Hg, diastolic BP > 100 mm Hg. Individuals with a history of hypertension may be allowed to participate in the study if the study physician or medical provider determines that the condition is stable and will not jeopardize the individual's safety.
* Hypotension (with symptoms) - systolic BP < 90 mm Hg, diastolic BP < 60 mm Hg.
* Coronary heart disease with symptoms (e.g., chest pain)
* Heart attack in the past year
* Cardiac rhythm disorder (irregular heart rhythm with symptoms)
* Chest pain in the last month (unless history indicates a non-cardiac source)
* Symptomatic heart disorder such as heart failure
* Advanced liver or kidney disease that requires medication or dialysis, paracentesis
* Major gastrointestinal illness (e.g. Celiac disease, Crohn's dx Ulcerative Colitis)
* Bleeding stomach ulcers in the past 30 days
* Lung disease that requires oxygen
* Major brain disorder (including stroke with residual deficit, brain tumor, and seizure disorder)
* Migraine headaches that occur more frequently than once per week
* Recent, unexplained fainting spells
* Problems giving blood samples
* Diabetes with insulin use or with HbA1C over 7%
* Current cancer or treatment for cancer in the past six months (except basal or squa-mous cell skin cancer)
* HIV, Hepatitis B, or Hepatitis C
* History of Tuberculosis or recent positive purified protein derivative (PPD)
* Other major medical condition (as determined by study physician)
* Currently symptomatic psychiatric disease (as determined by study physician)
* Psychosis, bipolar disorder, or psychiatric hospitalization within the past 12 months
* Suicidal ideation (thinking about ways to commit suicide) (within the past 12 months) or a lifetime occurrence of attempted suicide;
* Current depression - The Patient Health Questionnaire PHQ-9 for Depression will be used to screen for current (within 2 weeks) depression. Potential subjects who score >9 (or who score >0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way") will be excluded from study participation, and, at the discretion of the study physician, referred to appropriate psychiatric treatment;
* Pregnant or nursing mothers
* Use (within the past 30 days) of:

  * Illegal drugs (or if the urine drug screen is positive for tetrahydrocannabinol (THC), Cocaine, Amphetamine, Opiates, Methamphetamines, phencyclidine (PCP), Benzodiazepines, or Barbiturates), unless recent use of prescription Opiates or Benzodiazepines were taken for management of acute symptoms (e.g., tooth extraction, recent surgery);
  * Experimental (investigational) drugs;
  * Psychiatric medications including antidepressants (selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressant (TCAs), monoamine oxidase inhibitors (MAOIs), St. John's Wort), lithium, anti-psychotics or any other medications that are known to affect smoking cessation (e.g. clonidine);
  * Phentermine, triptans, tryptophan, linezolid, dextromethorphan, opiates (unless taken for management of acute symptoms), tramadol, or dopamine agonists;
  * Any agents that have documented correlation with increased incidence of valvulopathy and/or pulmonary hypertension (e.g., cyproheptadine, trazodone, nefazodone, amoxapine, tricyclic antidepressants, mirtazapine, pergolide, ergotamine, methysergide) (or anticipated use during the study);
  * Wellbutrin, bupropion, Zyban, Chantix, varenicline, nicotine patch, nicotine replacement therapy or any other smoking cessation aid;
  * Use of cigars, cigarillos, pipes, Hookah, dissolvable nicotine, snuff, chewing tobacco, or e-cigarettes
* Concurrent use of a serotonergic agent/combination associated with severe serotonin syndrome (within the past 30 days)
* Use of cigars, cigarillos, pipes, Hookah, dissolvable nicotine, snuff, chewing tobacco, or e-cigarettes within the past 30 days
* Self-report of consuming more than 6 alcoholic drinks on 1 or more days per week
* Significant adverse reaction to nicotine patch in the past
* Current participation or recent participation (in the past 30 days) in another smoking study at our Center or another research facility
* Current participation in another research study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed E. Rose, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke Center for Smoking Cessation, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicotine E-cigs + Nicotine Patches | Non-nicotine E-cigs + Nicotine Patches | Nicotine E-cigs + Placebo Patches | Non-nicotine E-cigs + Placebo Patches
Started | 37 | 33 | 11 | 13
Completed | 26 | 19 | 7 | 10
Not Completed | 11 | 14 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine E-cigs + Nicotine Patches | Non-nicotine E-cigs + Nicotine Patches | Nicotine E-cigs + Placebo Patches | Non-nicotine E-cigs + Placebo Patches | Total
Number analyzed (Participants) | 37 | 33 | 11 | 13 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (9.4) | 46.0 (8.7) | 46.3 (12.5) | 45.4 (8.7) | 47.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 17 | 6 | 8 | 56
  Male | 12 | 16 | 5 | 5 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 37 | 33 | 11 | 13 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 7 | 5 | 7 | 28
  White | 25 | 23 | 6 | 6 | 60
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 33 | 11 | 13 | 94
Baseline expired air carbon monoxide level [Mean (Standard Deviation); unit: Parts per million (ppm)] | 30.2 (14.3) | 27.7 (14.0) | 27.2 (13.4) | 28.5 (10.7) | 28.7 (13.5)

OUTCOME MEASURES:

1. Primary Outcome: Expired Air Carbon Monoxide (CO) to Assess Recent Smoking
Description: The effects of e-cigarette nicotine content and patch nicotine content on the concurrent use of conventional cigarettes will be assessed by comparing the groups on the expired air carbon monoxide (CO) measured at the end of the exposure period (Week 8).
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: Parts per million (ppm)
Arm/Group | Nicotine E-cigs + Nicotine Patches | Non-nicotine E-cigs + Nicotine Patches | Nicotine E-cigs + Placebo Patches | Non-nicotine E-cigs + Placebo Patches
Number analyzed (Participants) | 26 | 19 | 7 | 10
Parts per million (ppm) | 18.3 (16.2) | 22.9 (12.6) | 21.3 (25.7) | 25.6 (16.6)
Statistical Analysis 1: Comparison: Nicotine E-cigs + Nicotine Patches vs Non-nicotine E-cigs + Nicotine Patches; Due to time and budget constraints a blinded decision was made and approved by the funding agency to limit further enrollment to the two conditions that provided nicotine patches. The primary (one-tailed) test compared Nicotine e-cigs + Nicotine patches to Non-nicotine e-cigs + Nicotine patches; Test type: Superiority; p = 0.01, Regression, Linear

2. Secondary Outcome: Cigarette Use, Assessed by Self-report in Daily Dairies
Description: The effects of e-cigarette nicotine content and patch nicotine content on the concurrent use of conventional cigarettes will be assessed by comparing the groups on self-report of cigarette consumption on daily diaries (for week 8 only, average cigarettes smoked per day).
Time Frame: Week 8
Population: Participants with data available at week 8.
Measure: Mean (Standard Deviation); unit: cigarettes smoked per day
Arm/Group | Nicotine E-cigs + Nicotine Patches | Non-nicotine E-cigs + Nicotine Patches | Nicotine E-cigs + Placebo Patches | Non-nicotine E-cigs + Placebo Patches
Number analyzed (Participants) | 27 | 22 | 7 | 10
cigarettes smoked per day | 9.2 (7.7) | 9.9 (9.0) | 10.3 (12.3) | 9.3 (6.9)
Statistical Analysis 1: Comparison: Nicotine E-cigs + Nicotine Patches vs Non-nicotine E-cigs + Nicotine Patches; Test type: Superiority; p = 0.8, ANOVA

3. Secondary Outcome: E-cigarette Use, Assessed by Self-report in Daily Dairies
Description: The effects of e-cigarette nicotine content and patch nicotine content on the concurrent use of e-cigarettes will be assessed by comparing the groups on self-report of e-cigarette use on daily diaries (for week 8 only).
Time Frame: Week 8
Population: Participants with data available at week 8.
Measure: Mean (Standard Deviation); unit: e-cigarette pods per day
Arm/Group | Nicotine E-cigs + Nicotine Patches | Non-nicotine E-cigs + Nicotine Patches | Nicotine E-cigs + Placebo Patches | Non-nicotine E-cigs + Placebo Patches
Number analyzed (Participants) | 25 | 18 | 7 | 10
e-cigarette pods per day | 2.5 (2.6) | 2.0 (2.5) | 3.5 (3.6) | 2.4 (2.1)
Statistical Analysis 1: Comparison: Nicotine E-cigs + Nicotine Patches vs Non-nicotine E-cigs + Nicotine Patches; Test type: Superiority; p = 0.5, ANOVA

4. Secondary Outcome: Total Urinary 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL)
Description: The effects of e-cigarette nicotine content and patch nicotine content on the concurrent use of conventional cigarettes will be assessed by comparing the groups on total urinary NNAL, a metabolite of the tobacco-specific carcinogen 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK), at the end of week 8.
Time Frame: Week 8
Population: Data not collected due to time and budgetary limitations.
Arm/Group | Nicotine E-cigs + Nicotine Patches | Non-nicotine E-cigs + Nicotine Patches | Nicotine E-cigs + Placebo Patches | Non-nicotine E-cigs + Placebo Patches
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Adverse events were assessed through systematic approach. Solicited events were tabulated by asking participants to report side effects potentially common in e-cigarette use (e.g. throat irritation) and nicotine patch use (e.g. skin redness). Additionally, unsolicited events were tabulated by asking participants to report on any health concern that may have occurred during the study.
Arm/Group | Nicotine E-cigs + Nicotine Patches | Non-nicotine E-cigs + Nicotine Patches | Nicotine E-cigs + Placebo Patches | Non-nicotine E-cigs + Placebo Patches
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/33 | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/37 | 3/33 | 1/11 | 0/13
Other Adverse Events (participants affected / at risk) | 21/37 | 15/33 | 4/11 | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine E-cigs + Nicotine Patches (N=37) | Non-nicotine E-cigs + Nicotine Patches (N=33) | Nicotine E-cigs + Placebo Patches (N=11) | Non-nicotine E-cigs + Placebo Patches (N=13)
Knee Surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Knee arthritis resulted in knee instability resulted in fall resulted in knee surgery required hospitalization. Medical determination: not study related.
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Recurrent COPD exacerbation with hospitalization. The participant had two COPD exacerbations within 9 months of starting the study and 1 COPD exacerbation during study, but prior to initiating product use. Medical determination: not study related.
Infected renal stone (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Infected renal stones requiring hospitalization. Medical determination: not study related.
Streptococcal Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Strep throat resulted in likely streptococcal pneumonia with hospitalization. Medical determination: not study related.
Auditory Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Poly-substance use with caffeine, THC, kava kava, alcohol and kratom resulted in auditory hallucinations requiring hospitalization. Medical determination: not study related.
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hypertensive crisis (BP 245/130) occurred in a patient with a history of hypertension and resolved after treatment in the emergency room. Medical determination: not study related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotine E-cigs + Nicotine Patches (N=37) | Non-nicotine E-cigs + Nicotine Patches (N=33) | Nicotine E-cigs + Placebo Patches (N=11) | Non-nicotine E-cigs + Placebo Patches (N=13)
Headache (Nervous system disorders) | 2 | 0 | 1 | 0
Dizziness (Vascular disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 0 | 0
Insomnia (General disorders) | 0 | 3 | 0 | 1
Vivid Dreams (General disorders) | 7 | 6 | 3 | 1
Dry Mouth (General disorders) | 2 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Rapid Heart Beat (Cardiac disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Itchiness (Skin and subcutaneous tissue disorders) | 8 | 3 | 1 | 1 — Itchiness at the site of the nicotine or placebo patch
Irritability (Psychiatric disorders) | 2 | 2 | 1 | 0
Local Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 — Rash at site of nicotine or placebo patch
Distant Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 — Rash not at the site of the nicotine or placebo patch
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Version 1 (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT03492463/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Version 2 (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT03492463/Prot_SAP_001.pdf